CLINICAL TRIAL: NCT01207427
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Evaluate the Efficacy and Safety of ADL5945 for the Treatment of Opioid-induced Constipation in Adults Taking Opioid Therapy for Chronic Noncancer Pain
Brief Title: Evaluation of the Efficacy and Safety of ADL5945 for the Treatment of Opioid-induced Constipation in Adults Taking Opioid Therapy for Chronic Noncancer Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2402-001; 45CL242 (Other: Cubist Study Number)
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Opioid Induced Constipation
Keywords: opioid therapy; constipation; chronic noncancer pain; mu opioid receptor antagonist; ADL5945
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Each participant received 1 placebo capsule orally twice daily (BID) during the Run-in Placebo Period (1 week), the Double-blind Treatment Period (4 weeks), and the Run-out Placebo Period (1 week).
  Interventions: Drug: Placebo
- ADL5945 0.1 mg (Experimental): During the Run-in Placebo Period, each participant received 1 placebo capsule orally BID for 1 week. Then during the Double-blind Treatment Period, each participant received one 0.1-milligrams (mg) ADL5945 capsule orally BID for 4 weeks. Then during the Run-out Placebo Period, each participant received 1 placebo capsule orally BID for 1 week.
  Interventions: Drug: Placebo; Drug: ADL5945 0.1 mg
- ADL5945 0.25 mg (Experimental): During the Run-in Placebo Period, each participant received 1 placebo capsule orally BID for 1 week. Then during the Double-blind Treatment Period, each participant received one 0.25-mg ADL5945 capsule orally BID for 4 weeks. Then during the Run-out Placebo Period, each participant received 1 placebo capsule orally BID for 1 week.
  Interventions: Drug: Placebo; Drug: ADL5945 0.25 mg

INTERVENTIONS:
Drug: Placebo
Drug: ADL5945 0.1 mg
  Arms: ADL5945 0.1 mg
Drug: ADL5945 0.25 mg
  Arms: ADL5945 0.25 mg

SUMMARY:
Morphine and related opioid analgesics are known to slow gastrointestinal (GI) motility and reduce intestinal secretion through their binding to μ opioid receptors (MORs) within the GI tract. The most common symptoms associated with the effects of opioids are constipation and nausea and/or vomiting. Moreover, constipation is a common and distressing side effect of long-term opioid therapy.

The primary objective of this study was to compare ADL5945, a MOR antagonist, with placebo in the treatment of opioid-induced constipation (OIC) in adults taking long-term opioid therapy for chronic noncancer pain.

ELIGIBILITY:
Key Inclusion Criteria

* be a man or woman aged 18 to 75 years, inclusive, at the time of screening
* have a body weight ≥45 kilograms (kg) and a body mass index (BMI) ≤40 kilograms per square meter (kg/m^2)
* be taking a stable daily dose of opioids of ≥30-milligrams (mg) morphine-equivalent total -daily dose for chronic noncancer pain for ≥30 days before screening
* have opioid-induced constipation (OIC) by history. Additionally, based on the data collected during the 1-week screening period, participants must have <3 spontaneous bowel movements (SBMs) per week and have experienced ≥1 other bowel movement (BM) symptom (that is, straining to pass a stool, lumpy hard stools or small pellets, or sense of incomplete evacuation after passing a stool) for ≥25% of the total BMs
* be willing to discontinue use of all laxatives and stool softeners during the study period except as allowed by the protocol

Key Exclusion Criteria

* be pregnant, lactating, or planning to become pregnant during the study
* have aspartate aminotransferase (AST), alanine aminotransferase (ALT), blood urea nitrogen, or serum creatinine results ≥ 2 times the upper limit of normal
* have a recent history of myocardial infarction (MI) or unstable angina
* have an active malignancy of any type
* be taking opioids primarily for fibromyalgia
* be taking methadone as a maintenance medication (participants taking methadone for pain may be enrolled)
* be taking intrathecal opioids for the management of pain
* be taking tramadol, tapentadol, or any mixed agonist/antagonist opioid analgesics as the sole opioid for analgesia
* be taking any μ-opioid receptors (MOR) antagonist, including opioids in combination with naloxone, naltrexone, or methylnaltrexone bromide
* be taking medical marijuana for pain
* have gastrointestinal (GI) or pelvic disorders known to affect bowel transit, produce GI obstruction, or contribute to bowel dysfunction
* have taken antispasmodics, antidiarrheals, or prokinetics within 7 days before the start of the screening week
* be taking nonopioid medications known to cause constipation
* be taking antidiarrheals and have an incidence or a history of intermittent diarrhea or loose stools
* be unwilling to abstain from grapefruit and grapefruit-containing products
* have a history of alcoholism or illicit drug dependence or abuse within 5 years before screening
* have positive results on a urine drug screen (excluding opioids) that indicate illicit drug use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-10-14 (Actual); Primary Completion 2011-04-18 (Actual); Study Completion 2011-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Berger, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Run-in Placebo Period
Arm/Group | ADL5945 0.1 mg | ADL5945 0.25 mg | Placebo
Started | 43 | 45 | 43
Completed | 43 | 45 | 43
Not Completed | 0 | 0 | 0
Period: Double-blind Treatment Period
Arm/Group | ADL5945 0.1 mg | ADL5945 0.25 mg | Placebo
Started | 43 | 45 | 43
Received at Least 1 Dose of Study Drug | 43 | 45 | 43
Completed | 40 | 43 | 41
Not Completed | 3 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Run-out Placebo Period
Arm/Group | ADL5945 0.1 mg | ADL5945 0.25 mg | Placebo
Started | 40 | 43 | 41
Completed | 40 | 43 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- ADL5945 0.1 mg: During the Run-in Placebo Period, each participant received 1 placebo capsule orally BID for 1 week. Then during the Double-blind Treatment Period, each participant received one 0.1 mg ADL5945 capsule orally BID for 4 weeks. Then during the Run-out Placebo Period, each participant received 1 placebo capsule orally BID for 1 week.
- Total: Total of all reporting groups
Arm/Group | ADL5945 0.1 mg | ADL5945 0.25 mg | Placebo | Total
Number analyzed (Participants) | 43 | 45 | 43 | 131
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0 | 0 | 0 | 0
  BTWN | 40 | 44 | 40 | 124
  GTE65 | 3 | 1 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 23 | 63
  Male | 23 | 25 | 20 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Average of Spontaneous Bowel Movements (SBMs) During Treatment
Description: An SBM was defined as a bowel movement (BM) with no laxative use in the previous 24 hours. Each weekly SBM average was calculated as follows: (7 × number of SBMs) / (number of days with nonmissing data). The overall SBM rate for the 4-week double-blind treatment period was calculated as follows: (the average of the first week + the average of the second week + the average of the third week + the average of the fourth week) / 4.
Time Frame: Baseline, Weeks 1 through 4 of treatment
Population: All participants who were randomized to study treatment and had at least 1 evaluable SBM post-dose measurement during the Double-blind Period. Last-observation-carried-forward (LOCF) was used to impute missing postbaseline values.
Measure: Mean (Standard Error); unit: Number of SBMs/week
Groups:
- ADL5945 0.1 mg: During the Run-in Placebo Period, each participant received 1 placebo capsule orally BID for 1 week. Then during the Double-blind Treatment Period, each participant received one 0.1-mg ADL5945 capsule orally BID for 4 weeks. Then during the Run-out Placebo Period, each participant received 1 placebo capsule orally BID for 1 week.
Arm/Group | ADL5945 0.1 mg | ADL5945 0.25 mg | Placebo
Number analyzed (Participants) | 43 | 45 | 43
Number of SBMs/week | 1.96 (0.35) | 3.42 (0.49) | 1.44 (0.27)

ADVERSE EVENTS:
Groups:
- ADL5945 0.1 mg: During the Run-in Placebo Period, each participant received 1 placebo capsule orally BID for 1 week. Then during the Double-blind Treatment Period, each participant received one 0.1- mg ADL5945 capsule orally BID for 4 weeks. Then during the Run-out Placebo Period, each participant received 1 placebo capsule orally BID for 1 week.
Arm/Group | ADL5945 0.1 mg | ADL5945 0.25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/43 | 2/45 | 0/43
Other Adverse Events (participants affected / at risk) | 14/43 | 19/45 | 15/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADL5945 0.1 mg (N=43) | ADL5945 0.25 mg (N=45) | Placebo (N=43)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ADL5945 0.1 mg (N=43) | ADL5945 0.25 mg (N=45) | Placebo (N=43)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Oral Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Adverse Drug Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug Withdrawal Syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 5 (5) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0/20 (0) | 1/20 (1) | 0/23 (0)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Burns First Degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other